Treatment of HFpEF with nitrate supplement: A double-blind, placebo controlled trial including patients with atrial fibrillation

Principal Investigator: Ralph Hamill, MD

NCT #03289481

Document date: March 20, 2019

A t-test was utilized to examine the difference between the change in outcome measures for the exercise echocardiogram: diastolic dysfunction (E/E'), estimated right ventricular systolic pressure (TR), metabolic equivalents (METS), and time on the treadmill among the treatment and the placebo groups. The change in outcome measures were calculated by subtracting the pre-stress test measure from the post-stress test measure at the time of the patient encounter. T-values were considered significant at the .05 level. Analysis was done using SAS Enterprise Guide 7.1.

Document date: March 20, 2019